CLINICAL TRIAL: NCT03842891
Title: Genetic Variants Modulate Association Between Dietary n-3 LCPUFAs and DHA Proportion in Breast Milk
Status: Completed | Type: Observational
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMUH106-REC1-115
Record Dates: First submitted 2019-02-14; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Fatty Acid Desaturases; Polymorphism, Single Nucleotide; Milk, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
DHA is important for the development of brain and retina in newborns. Considering that exclusive breast feeding for at least 4 ~6 months are globally recommended, plus it is well known that nutrient requirement is determined by both genetic and environmental (including diet) factors, this clinical study sought to investigate how the DHA levels in maternal milk is modulated by genetic variants and dietary n-3 LCPUFA intake. To recruit subjects (n=193), the inclusion criteria are Han Chinese women just having delivered full-term baby, 20-40 years old, healthy, and willing to breast feed their baby for at least 2 months. Written informed consent will be obtained from participants. Personal information (or covariates) such as height, weight (before getting pregnancy and delivery, respectively), age, parity, education, smoking, alcohol drinking, gender of baby…etc, and DNA from oral swab will be collected. Breast milk and dietary data will be collected at the end of the 1st and 2nd month of postpartum period. Considering Han Chinese women usually have special postpartum diets and care during puerperium, therefore, collection of breast milk and dietary information will be repeated at the 2nd month. The fatty acid composition in milk will be analyzed by gas chromatography. Using food frequency questionnaire, intake of n-3 LCPUFA from foods + fish oil supplements will be calculated. Subjects will be instructed to give a 3-days food record as well. We foresee results of this study might contribute to public health care as nutritionists/dietitians will be able to target the vulnerable subjects, who are dietary dependent for DHA, for dedications in nutrition consults or customized dietary guidance. Moreover, these information are valuable in making policy regarding dietary recommendation in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Han Chinese women
* Full-term pregnancy(>36weeks)
* 20-40 years old
* Healthy
* Breast feed their baby for at least 2 months

Exclusion Criteria:

* Death before and after childbirth
* Child with congenital disease

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Of all 193 participants, there were 180 who continued to track for two months.
Sampling Method: Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2018-09-25 (Actual)

PRIMARY OUTCOMES:
Breast milk fatty acid composition | 2 month
  Breast milk will be collected at the end of the 1st and 2nd month of postpartum period.The fatty acid composition in milk will be analyzed by gas chromatography.

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Min Chao, PhD, Principal Investigator — China Medical University, China
Locations (1):
- China Medical University, Taichung, Taiwan

REFERENCES:
- [Derived] Wu WC, Lin HC, Liao WL, Tsai YY, Chen AC, Chen HC, Lin HY, Liao LN, Chao PM. FADS Genetic Variants in Taiwanese Modify Association of DHA Intake and Its Proportions in Human Milk. Nutrients. 2020 Feb 20;12(2):543. doi: 10.3390/nu12020543. PMID 32093185